CLINICAL TRIAL: NCT02079363
Title: Cell-free DNA Promoter Hypermethylation in Plasma From Patients With Pancreatic Adenocarcinoma, Compared to Patients With Pancreatitis and Pancreatitis and Patients Screened for, But Not Having Pancreatic Adenocarcinoma."
Brief Title: DNA Promoter Hypermethylation as a Blood Based Maker for Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, MD, DMSc, Consultant surgeant, Professor of Surgery, Aalborg University Hospital
Other Study IDs: Hypmet
Record Dates: First submitted 2014-03-04; First posted 2014-03-05 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Pancreatic Diseases; Pancreatic Neoplasms; Pancreatitis
Keywords: Pancreatic Diseases; Pancreatic Neoplasms; Pancreatitis; DNA promoter hypermethylation; DNA methylation; Cell-free DNA; Plasma
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Neoplasms; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell free methylated DNA in EDTA plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Patients with pancreatic adenocarcinoma: Exclusion criteria:
  No prior cancer. No anticoagulant treatment.
  Interventions: Other: No interventions, this is an observational study
- Patients with chronic pancreatitis: Exclusion criteria:
  No prior cancer. No anticoagulant treatment.
  Interventions: Other: No interventions, this is an observational study
- Patients with acute pancreatitis: Exclusion criteria:
  No prior cancer.
  Interventions: Other: No interventions, this is an observational study
- Patients screened for but not having upper GI cancer: Exclusion criteria:
  No prior cancer.
  Interventions: Other: No interventions, this is an observational study

INTERVENTIONS:
Other: No interventions, this is an observational study

SUMMARY:
The objectives of this project are to test whether alteration in DNA hypermethylation in plasma is:

* a diagnostic marker for pancreatic cancer
* a prognostic marker for pancreatic cancer
* a marker for recurrence of pancreatic cancer
* changing during the course of chronic pancreatitis, with the purpose of finding patients with high risk of developing pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic cancer (PCa) is one of the most deadly cancers with a 5-year survival rate of less than 10 %. The majority of PCa are found to be none-resectable at the time of diagnosis. Only 10 - 20% of patients are offered surgical treatment, which is the only chance of cure. The mean survival times of none-resected patients are 3 to 6 months. Despite surgical treatment many patients experience recurrence. The high overall mortality is mainly caused by difficulties in early diagnosis due to unspecific/lack of symptoms in the early stages of the disease.

Patients with resectable tumors and no co-morbidity, have a 5-year survival rate up to 54 %. This indicates that early detection of the disease, which enables complete surgical resection of the tumor, is a way to improve survival. Chronic pancreatitis is one of the only known risk factors for PCa.

Currently there is no valid diagnostic marker for PCa. Diagnosis requires advanced methods and several of these are invasive and entail a risk of complications. A blood-based marker for pancreatic cancer would be a major achievement and of great benefit to the patients, and may even be used in screening.

During development of cancer changes in DNA arise, including DNA hypermethylation where a methyl residue is attached to the DNA. The methylation most frequently occurs in the regulatory region of the gene leading to inactivity. Some of the inactivated genes are necessary to ensure the control of cell growth. When these genes are inactivated, the cell will no longer be subject to normal control mechanisms and may eventually develop into a cancer cell.

Small amounts of DNA are released into the blood and can be detected in a blood sample. The DNA changes may be tumor specific and potentially useable as a marker for PCa. In 2012 our research unit in cooperation with Department of Molecular Diagnostic, Aalborg University Hospital published an optimized method for detection of hypermethylated DNA in plasma. The method has greatly improved sensitivity.

The purpose of our study is to test whether alterations in DNA hypermethylations in blood can be used as:

* A diagnostic marker for pancreatic cancer.
* A prognostic marker for pancreatic cancer.
* A marker for recurrence.
* Monitoring patients with chronic pancreatitis and detecting patients with particularly high risk of developing pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pancreatitis who are hospitalized or have an outpatient visit at Aalborg University Hospital Or
* Patients hospitalized at Aalborg University Hospital, with acute pancreatitis verified by UL, CT or MR-scan and/or increased s-amylase

Exclusion Criteria:

* Prior cancer history.
* Anticoagulant therapy.
* Immunological tissue disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic adenocarcinoma, who were referred to Aalborg University Hospital between 2008 and 2012. Blodsamples are stored in a biobank.
  Patients with chronic pancreatitis, who are hospitalized or have an outpatient visit at Aalborg University Hospital.
  Patients with acute pancreatitis, who are hospitalized at Aalborg University Hospital.
  Patients who are referred to Aalborg University Hospital for suspected upper GI cancer. Subsequent examinations invalidate the cancer diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of methylated genes for each participant. | Time of diagnosis
  We investigate the methylation status a of panel of 20 different genes in cell-free DNA in plasma. Plasma from patients with c. pancreas will be compared to plasma from patients in the control groups to se if DNA promoter hypermethylation can be used as a diagnostic marker for pancreas cancer.

SECONDARY OUTCOMES:
Number of methylated genes for each participant related to prognosis | 2 years follow up
  We investigate the methylation status a of panel of 20 different genes in cell-free DNA in plasma. Number of methylated genes will be investigated in relation to TNM- classification, tumor-size and time of survival.

OTHER OUTCOMES:
Number of methylated genes in patients who are undergoing curative surgery. | 2 years follow up
  We investigate the methylation status a of panel of 20 different genes in cell-free DNA in plasma from patients diagnosed with c. pancreas before curative surgery and after surgery and every 3 months for a 2 years periode. The purpose is to study the methylation status as a marker of recurrence.
Number of methylated genes in patients with chronic pancreatitis. | 2 years follow up
  We investigate the methylation status a of panel of 20 different genes in cell-free DNA in plasma form patients with chronic pancreatitis. The purpose is to se if the methylation profile changes during the course of chronic pancreatitis and to detect chronic pancreatitis patients with particular high risk of developing pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Stine Dam Henriksen, MD, Principal Investigator — Department of Gastrointestinal Surgery, Aalborg University Hospital, Denmark; Ole Thorlacius-Ussing, MD,DMSc,Prof, Study Chair — Department of Gastrointestinal Surgery, Aalborg University Hospital, Denmark
Locations (1):
- Research unit, Surgical Department of Gastroenterology, Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Background] Park JW, Baek IH, Kim YT. Preliminary study analyzing the methylated genes in the plasma of patients with pancreatic cancer. Scand J Surg. 2012;101(1):38-44. doi: 10.1177/145749691210100108. PMID 22414467
- [Background] Melson J, Li Y, Cassinotti E, Melnikov A, Boni L, Ai J, Greenspan M, Mobarhan S, Levenson V, Deng Y. Commonality and differences of methylation signatures in the plasma of patients with pancreatic cancer and colorectal cancer. Int J Cancer. 2014 Jun 1;134(11):2656-62. doi: 10.1002/ijc.28593. Epub 2013 Nov 29. PMID 24288256
- [Background] Park JK, Ryu JK, Yoon WJ, Lee SH, Lee GY, Jeong KS, Kim YT, Yoon YB. The role of quantitative NPTX2 hypermethylation as a novel serum diagnostic marker in pancreatic cancer. Pancreas. 2012 Jan;41(1):95-101. doi: 10.1097/MPA.0b013e318221c903. PMID 21778928
- [Background] Liggett T, Melnikov A, Yi QL, Replogle C, Brand R, Kaul K, Talamonti M, Abrams RA, Levenson V. Differential methylation of cell-free circulating DNA among patients with pancreatic cancer versus chronic pancreatitis. Cancer. 2010 Apr 1;116(7):1674-80. doi: 10.1002/cncr.24893. PMID 20143430
- [Background] Jiao L, Zhu J, Hassan MM, Evans DB, Abbruzzese JL, Li D. K-ras mutation and p16 and preproenkephalin promoter hypermethylation in plasma DNA of pancreatic cancer patients: in relation to cigarette smoking. Pancreas. 2007 Jan;34(1):55-62. doi: 10.1097/01.mpa.0000246665.68869.d4. PMID 17198183
- [Background] Yi JM, Guzzetta AA, Bailey VJ, Downing SR, Van Neste L, Chiappinelli KB, Keeley BP, Stark A, Herrera A, Wolfgang C, Pappou EP, Iacobuzio-Donahue CA, Goggins MG, Herman JG, Wang TH, Baylin SB, Ahuja N. Novel methylation biomarker panel for the early detection of pancreatic cancer. Clin Cancer Res. 2013 Dec 1;19(23):6544-6555. doi: 10.1158/1078-0432.CCR-12-3224. Epub 2013 Oct 2. PMID 24088737
- [Derived] Henriksen SD, Madsen PH, Larsen AC, Johansen MB, Drewes AM, Pedersen IS, Krarup H, Thorlacius-Ussing O. Cell-free DNA promoter hypermethylation in plasma as a diagnostic marker for pancreatic adenocarcinoma. Clin Epigenetics. 2016 Nov 16;8:117. doi: 10.1186/s13148-016-0286-2. eCollection 2016. PMID 27891190